CLINICAL TRIAL: NCT06822647
Title: Optimal Timing of Routine Cervical Length Measurements During Anatomy Survey
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Raminder Khangura, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16839
Record Dates: First submitted 2025-01-29; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Cervical Insufficiency; Preterm Birth; Cervical Length Measurement
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth

STUDY DESIGN:
Intervention Model Description: Participants are randomized to have cervical length measurements taken either at the beginning or the end of the anatomy survey.
Masking Description: No additional masking is used as this is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beginning of Anatomy Survey (Experimental): Participants in this arm will undergo cervical length measurement via transvaginal ultrasound at the start of the fetal anatomy survey. This timing aims to evaluate whether early measurement improves adherence to the nine CLEAR criteria for accurate cervical length assessment. Measurements will also be conducted using grayscale and sepia-filtered ultrasound imaging.
  Interventions: Procedure: Cervical Length Measurement at the Beginning of the Anatomy Survey
- End of Anatomy Survey (Experimental): Participants in this arm will undergo cervical length measurement via transvaginal ultrasound at the end of the fetal anatomy survey. This timing aims to evaluate whether late measurement improves adherence to the nine CLEAR criteria for accurate cervical length assessment. Measurements will also be conducted using grayscale and sepia-filtered ultrasound imaging.
  Interventions: Procedure: Cervical Length Measurement at the End of the Anatomy Survey

INTERVENTIONS:
Procedure: Cervical Length Measurement at the Beginning of the Anatomy Survey — This intervention involves performing a transvaginal ultrasound to measure cervical length at the beginning of the fetal anatomy survey. The procedure includes using both grayscale and sepia-filtered imaging to evaluate adherence to the nine CLEAR criteria for accurate cervical length assessment.
  Arms: Beginning of Anatomy Survey
Procedure: Cervical Length Measurement at the End of the Anatomy Survey — This intervention involves performing a transvaginal ultrasound to measure cervical length at the end of the fetal anatomy survey. The procedure includes using both grayscale and sepia-filtered imaging to evaluate adherence to the nine CLEAR criteria for accurate cervical length assessment.
  Arms: End of Anatomy Survey

SUMMARY:
The goal of this clinical trial is to determine the optimal timing for measuring cervical length (CL) during fetal anatomy surveys in pregnant individuals. This study focuses on improving the accuracy of cervical length assessments, which are critical for identifying individuals at risk for preterm birth. The main questions it aims to answer are:

* Does measuring cervical length at the beginning of the anatomy survey result in a higher proportion of scans meeting the nine CLEAR (Cervical Length Education and Review) criteria compared to measuring at the end of the survey?
* Does the use of sepia-filtered ultrasound images improve the proportion of scans meeting the nine CLEAR criteria compared to conventional grayscale images?

Researchers will compare two groups of participants randomized to have cervical length measured either at the beginning or at the end of the anatomy survey. Additionally, all participants will undergo cervical length measurements using both grayscale and sepia-filtered ultrasound imaging.

Participants will:

* Receive a patient information sheet through MyChart explaining the study and standard cervical length screening during anatomy surveys.
* Provide verbal consent for a transvaginal ultrasound and study participation.
* Be randomized to have their cervical length measured at either the start or end of the fetal survey.
* Undergo cervical length measurement using both grayscale and sepia-filtered ultrasound imaging modalities.
* This study involves no additional risks beyond those of routine clinical care and aims to enhance clinical practice by identifying optimal methods for cervical length assessment during pregnancy.

DETAILED DESCRIPTION:
Study Title: Optimal Timing of Routine Cervical Length Measurements During Anatomy Survey

Study Aim and Background: This randomized controlled trial investigates whether the timing of cervical length measurements during fetal anatomy surveys impacts the accuracy of assessments. Current guidelines recommend transvaginal cervical length screening during anatomy surveys to identify individuals at risk for preterm birth. However, the guidelines do not specify whether measurements should be taken at the beginning or end of the ultrasound exam, a lengthy procedure (60-90 minutes) that may introduce uterine contractions and distort results. Additionally, the study evaluates whether using sepia-filtered ultrasound images can enhance measurement accuracy compared to conventional grayscale imaging.

Primary Hypothesis: Cervical lengths measured at the beginning of the fetal survey will result in a higher proportion of scans meeting the nine CLEAR criteria than those measured at the end.

Secondary Hypothesis: Sepia-filtered ultrasound imaging will yield a greater proportion of scans meeting the CLEAR criteria compared to grayscale imaging.

Study Design:

* Type: Randomized controlled trial.
* Setting: Conducted across all Maternal Fetal Medicine (MFM) ultrasound units within Henry Ford Health (HFH).
* Population: Pregnant individuals between 16w0d and 23w6d gestation undergoing fetal anatomy surveys. Participants with a history of preterm birth or cervical insufficiency are excluded.
* Intervention: Randomization of participants to have cervical length measurements taken at either the beginning or end of the anatomy survey. Measurements will be performed using both grayscale and sepia-filtered imaging modalities.
* Randomization: Pre-prepared envelopes (n=550) direct sonographers to perform cervical length measurement either at the start or end of the anatomy survey. Envelopes are indistinguishable and shuffled to ensure blinding.

Procedures:

Patient Enrollment:

* Prior to the anatomy scan, participants receive a MyChart information sheet outlining the study.
* Participants provide verbal consent for cervical length measurement via transvaginal ultrasound and for study participation.
* Verbal consent is documented in the patient's chart.

Randomization:

* Upon consent, the sonographer randomly selects an envelope to determine the timing of cervical length measurement.
* Cervical length measurements are conducted per routine care, ensuring the bladder is emptied beforehand.

Data Collection:

* Cervical length is measured using both grayscale and sepia-filtered ultrasound images.
* Sonographers save the first image with the word "CLEAR" to indicate study participation.
* MFM physicians complete a worksheet assessing the nine CLEAR criteria for each scan. These worksheets are de-identified and stored securely in a binder.

Data Security:

* Worksheets containing study data are stored in a secure MFM physician workroom, accessible only via HFH badge access.
* De-identified data is entered into a secure database, password-protected and accessible only to authorized personnel. The database will be erased following data analysis and publication.

Analysis Plan:

* Primary Analysis: Proportion of scans meeting the nine CLEAR criteria will be compared between groups (cervical length measured at beginning vs. end of survey) using chi-square tests. Logistic regression will adjust for confounders such as gestational age and sonographer experience.
* Secondary Analysis: Effect of sepia-filtered imaging on CLEAR criteria adherence will be evaluated using paired t-tests or Wilcoxon signed-rank tests. Interaction analysis will assess the combined effects of timing and imaging modality using two-way ANOVA or logistic regression.
* Handling Missing Data: Multiple imputation techniques will address missing values in the CLEAR criteria.
* Sample Size: A total of 550 participants (275 per group) provides 80% power to detect a 10-15% difference in the proportion of scans meeting the CLEAR criteria, assuming a baseline adherence of 60%.

Anticipated Risks and Benefits:

* Risks: No additional risks beyond standard cervical length screening.
* Benefits: Improved accuracy in cervical length measurements could optimize clinical decision-making and patient outcomes, particularly for managing short cervix during pregnancy.

Confidentiality:

* No personally identifiable information (PHI) is linked to study worksheets or data.
* IRB-approved procedures ensure confidentiality and data integrity.

Investigator Qualifications:

* Primary Author: Shelby Masters, MD, MFM Fellow.
* Principal Investigator: Raminder Khangura, MD, MFM Attending.
* Co-Investigators: Nicolina Smith, DO, and Shahd Karrar, MD, MFM Fellows.

This innovative study, which has not been explored previously in the literature, has the potential to influence clinical guidelines for cervical length measurement during pregnancy, ensuring more reliable assessments and improved care for at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals between 16 weeks and 23 weeks + 6 days of gestation.
* Presenting for a fetal anatomy survey at Henry Ford Health MFM ultrasound units.
* Consent to a transvaginal cervical length measurement as part of routine care.
* Agreement to participate in the study, including randomization for the timing of cervical length measurement.

Exclusion Criteria:

* History of preterm delivery.
* Diagnosis of cervical insufficiency.
* Declines or unable to consent to a transvaginal cervical length measurement.
* Patients receiving care at non-Henry Ford Health radiology clinics.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Cervical Length Measurements Meeting CLEAR Criteria at time of anatomy scan, between 18-24 weeks gestation, measured by transvaginal ultrasound | At the time of the fetal anatomy survey, specifically 18-24wks (one-time measurement per participant).
  The primary outcome is the proportion of transvaginal cervical length measurements that meet all nine CLEAR (Cervical Length Education and Review) criteria for accuracy. This will assess whether timing (beginning vs. end of anatomy survey) impacts measurement reliability.

SECONDARY OUTCOMES:
Proportion of Scans Meeting CLEAR Criteria Using Sepia-Filtered Imaging | At the time of the fetal anatomy survey, specifically 18-24wks (one-time measurement per participant).
  The secondary outcome evaluates whether sepia-filtered ultrasound imaging improves adherence to the nine CLEAR criteria compared to conventional grayscale imaging. Measurements will be analyzed for both imaging modalities.

OTHER OUTCOMES:
Interaction Between Timing and Imaging Modality on CLEAR Criteria Adherence | At the time of the fetal anatomy survey, specifically 18-24wks (one-time measurement per participant).
  This exploratory outcome examines whether the timing of cervical length measurement (beginning vs. end of the anatomy survey) interacts with the imaging modality (grayscale vs. sepia-filtered) to influence adherence to the nine CLEAR criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Raminder Khangura, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health New Center One, Detroit, Michigan, United States